CLINICAL TRIAL: NCT00390221
Title: Multicenter, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Determine the Safety and Efficacy of Daclizumab HYP (DAC HYP) as a Monotherapy Treatment in Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: Safety and Efficacy Study of Daclizumab High Yield Process (DAC HYP) to Treat Relapsing-Remitting Multiple Sclerosis
Acronym: SELECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 205-MS-201
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: MS; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — daclizumab HYP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive 3 subcutaneous (SC) injections of placebo every 4 weeks for up to 52 weeks.
  Interventions: Drug: Placebo
- 150 mg DAC HYP (Experimental): Participants will receive 3 SC injections every 4 weeks for up to 52 weeks.
  Interventions: Biological: BIIB019 (Daclizumab High Yield Process)
- 300 mg DAC HYP (Experimental): Participants will receive 3 SC injections every 4 weeks for up to 52 weeks.
  Interventions: Biological: BIIB019 (Daclizumab High Yield Process)

INTERVENTIONS:
Biological: BIIB019 (Daclizumab High Yield Process) — SC injection
  Other Names: DAC HYP; Daclizumab HYP
  Arms: 150 mg DAC HYP; 300 mg DAC HYP
Drug: Placebo — Placebo SC injection
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine whether DAC HYP, when compared to placebo, is effective in reducing the rate of relapses between baseline and Week 52. The secondary objectives are to determine whether DAC HYP is effective in reducing the number of new gadolinium (Gd)-enhancing lesions, reducing the number of new or newly-enlarging T2 hyperintense lesions, reducing the proportion of participants with relapses, and improving quality of life.

ELIGIBILITY:
Key Inclusion Criteria:

* Multiple Sclerosis (MS) subjects who have a confirmed diagnosis of relapsing-remitting MS according to McDonald criteria #1-4 and a baseline Expanded Disability Status Scale (EDSS) between 0.0 and 5.0, inclusive, who meet either of the following 2 criteria:

  * Have experienced at least 1 relapse within the 12 months prior to randomization, with a cranial magnetic resonance imaging (MRI) demonstrating lesion(s) consistent with MS , OR
  * Show evidence of gadolinium-enhancing lesions of the brain on an MRI performed within the 6 weeks prior to randomization.

Key Exclusion Criteria:

* Diagnosis of primary progressive, secondary progressive, or progressive relapsing MS
* History of malignancy
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity
* History of abnormal laboratory results based on investigator judgment
* History of human immunodeficiency virus (HIV) or other immunodeficient conditions
* History of drug or alcohol abuse within the 2 years prior to randomization
* An MS relapse that has occurred within the 50 days prior to randomization AND/OR the subject has not stabilized from a previous relapse prior to randomization
* Positive screening for active infection with Hepatitis B virus or Hepatitis C virus
* Varicella or herpes zoster virus infection or any severe viral infection within 6 weeks before Screening
* Exposure to varicella zoster virus within 21 days before Screening.
* Abnormal blood tests at Screening: Hemoglobin ≤9.0 g/dL, Platelets ≤100 × 10^9/L, Lymphocytes ≤1.0 × 10^9/L, Neutrophils ≤1.5 × 10^9/L, alanine aminotransferase/serum glutamate pyruvate transaminase (ALT/SGPT), aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT), or gamma-glutamyl-transferase >2 times the upper limit of normal (ULN) and serum creatinine >ULN.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 621 (Actual)
Dates: Start 2008-02; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (56):
- Czechia (4):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Pilsen
  - Research Site, Teplice
- Germany (5):
  - Research Site, Erlangen
  - Research Site, Marburg
  - Research Site, Osnabrück
  - Research Site, Regensburg
  - Research Site, Rostock
- Hungary (9):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Esztergom
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Siófok
  - Research Site, Zalaegerszeg
- India (7):
  - Research Site, Andra-Pradeash
  - Research Site, Bangalore
  - Research Site, Chennai
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, Rajasthan
  - Research Site, Visakhapatnam
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Warsaw
- Russia (11):
  - Research Site, Kazan'
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Smolensk
  - Research Site, Ufa
  - Research Site, Yaroslavl
- Ukraine (8):
  - Research Site, Chernivtsi
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Lviv
  - Research Site, Poltava
  - Research Site, Zaporizhzhya
- United Kingdom (5):
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Plymouth
  - Research Site, Sheffield
  - Research Site, Stoke-on-Trent

REFERENCES:
- [Derived] Huss DJ, Mehta DS, Sharma A, You X, Riester KA, Sheridan JP, Amaravadi LS, Elkins JS, Fontenot JD. In vivo maintenance of human regulatory T cells during CD25 blockade. J Immunol. 2015 Jan 1;194(1):84-92. doi: 10.4049/jimmunol.1402140. PMID 25416807
- [Derived] Gold R, Giovannoni G, Selmaj K, Havrdova E, Montalban X, Radue EW, Stefoski D, Robinson R, Riester K, Rana J, Elkins J, O'Neill G; SELECT study investigators. Daclizumab high-yield process in relapsing-remitting multiple sclerosis (SELECT): a randomised, double-blind, placebo-controlled trial. Lancet. 2013 Jun 22;381(9884):2167-75. doi: 10.1016/S0140-6736(12)62190-4. Epub 2013 Apr 4. PMID 23562009
- See also: (MSActiveSource.com is a resource for news, information, and disease management for all individuals touched by Multiple Sclerosis. This site is sponsored by Biogen Idec.) — http://www.msactivesource.com
- See also: (The website of the National Multiple Sclerosis Society, an organization dedicated to providing information to individuals with MS, their families, and healthcare providers.) — http://www.nationalmssociety.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo administered as 3 subcutaneous (SC) injections every 4 weeks for up to 52 weeks
- 150 mg DAC HYP: 150 mg Daclizumab High Yield Process (DAC HYP) administered as 3 SC injections every 4 weeks for up to 52 weeks
- 300 mg DAC HYP: 300 mg DAC HYP administered as 3 SC injections every 4 weeks for up to 52 weeks
Period: Overall Study
Arm/Group | Placebo | 150 mg DAC HYP | 300 mg DAC HYP
Started | 204 | 208 | 209
Completed | 186 | 188 | 194
Not Completed | 18 | 20 | 15
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Adverse Event | 1 | 4 | 3
Not completed — Investigator Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 13 | 9 | 7
Not completed — Subject Non-compliance | 1 | 0 | 2
Not completed — Other | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo administered as 3 SC injections every 4 weeks for up to 52 weeks
- 150 mg DAC HYP: 150 mg DAC HYP administered as 3 SC injections every 4 weeks for up to 52 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | 150 mg DAC HYP | 300 mg DAC HYP | Total
Number analyzed (Participants) | 204 | 208 | 209 | 621
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (9.02) | 35.3 (8.94) | 35.2 (8.67) | 35.7 (8.88)
Age, Customized [Number; unit: participants]
  18 to 19 years | 1 | 4 | 5 | 10
  20 to 29 years | 46 | 55 | 53 | 154
  30 to 39 years | 79 | 73 | 90 | 242
  40 to 49 years | 60 | 67 | 49 | 176
  50 to 55 years | 18 | 9 | 12 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 140 | 134 | 402
  Male | 76 | 68 | 75 | 219

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Annualized Relapse Rate Between Baseline and Week 52
Description: Relapses are defined as new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the examining neurologist. The annualized relapse rate was calculated as the total number of relapses that occurred during the study divided by the total number of subject-years followed in the study.
Time Frame: Baseline through Week 52
Population: Intent to treat population: all randomized participants who received at least 1 dose of study medication (excluding 21 participants from a single site due to a protocol violation in dosing).
Measure: Number (95% Confidence Interval); unit: relapses per person-years
Arm/Group | Placebo | 150 mg DAC HYP | 300 mg DAC HYP
Number analyzed (Participants) | 196 | 201 | 203
relapses per person-years | 0.458 [0.370 to 0.566] | 0.211 [0.155 to 0.287] | 0.230 [0.172 to 0.308]
Statistical Analysis 1: Comparison: Placebo vs 150 mg DAC HYP; Test type: Superiority or Other; p < 0.0001, Negative Binomial Regression — adjusted for the number of relapses in the 1 year prior to study entry, baseline Expanded Disability Status Scale (<=2.5 vs > 2.5), and age (<=35 vs >35); Rate Ratio = 0.461, 95% CI 2-sided [0.318 to 0.668]
Statistical Analysis 2: Comparison: Placebo vs 300 mg DAC HYP; Test type: Superiority or Other; p = 0.0002, Negative Binomial Regression — [p-value comment as in outcome 1, analysis 1]; Rate Ratio = 0.503, 95% CI 2-sided [0.352 to 0.721]

2. Secondary Outcome: Adjusted Mean Number of New Gadolinium (Gd)-Enhancing Lesions Between Week 8 and Week 24
Description: Gd-enhancing lesions are detected when Gd leaks into a perivascular space due to local breakdown of the blood-brain barrier, indicating the presence of active inflammation. For participants with missing data the last valid nonbaseline measurement was carried forward if the participant was missing only 1 or 2 consecutive postbaseline scans. Otherwise the mean based on treatment group and visit was used as the imputed value. Estimated from a negative binomial model adjusted for the baseline number of Gd-enhancing lesions.
Time Frame: Week 8 through Week 24
Population: Magnetic Resonance Imaging (MRI) Intensive Population: a protocol-defined subset of participants consisting of the first 307 participants enrolled in the study with non-missing baseline values.
Measure: Mean (95% Confidence Interval); unit: lesions
Arm/Group | Placebo | 150 mg DAC HYP | 300 mg DAC HYP
Number analyzed (Participants) | 104 | 101 | 102
lesions | 4.79 [3.56 to 6.43] | 1.46 [1.05 to 2.03] | 1.03 [0.73 to 1.46]
Statistical Analysis 1: Comparison: Placebo vs 300 mg DAC HYP; For each of the secondary endpoints, a sequential closed testing procedure was used, with the first comparison (the DAC HYP 300 mg group versus placebo) and the second comparison (the DAC HYP 150 mg group versus placebo). Secondary endpoints were rank prioritized, in the order presented. If statistical significance was not achieved for an endpoint, all endpoints(s) of a lower rank were not considered statistically significant; Test type: Superiority or Other; p < 0.0001, Negative Binomial Regression; adjusted for the baseline number of Gd-enhancing lesions; Percent Reduction = 78.44, 95% CI 2-sided [65.97 to 86.35]
Statistical Analysis 2: Comparison: Placebo vs 150 mg DAC HYP; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Negative Binomial Regression; adjusted for the baseline number of Gd-enhancing lesions; Percent Reduction = 69.47, 95% CI 2-sided [52.40 to 80.41]

3. Secondary Outcome: Adjusted Mean Number of New or Newly-enlarging T2 Hyperintense Lesions at Week 52
Description: Lesions detected on T2-weighted sequences represent a range of histopathology related to MS, including edema, inflammation, demyelination, gliosis, and axon loss.
Time Frame: Week 52
Population: Intent to treat population: all randomized subjects who received at least 1 dose of study medication (excluding 21 subjects from a single site due to a protocol violation in dosing) with a non-missing value at baseline.
Measure: Mean (95% Confidence Interval); unit: lesions
Arm/Group | Placebo | 150 mg DAC HYP | 300 mg DAC HYP
Number analyzed (Participants) | 195 | 199 | 200
lesions | 8.13 [6.65 to 9.94] | 2.42 [1.96 to 2.99] | 1.73 [1.39 to 2.15]
Statistical Analysis 1: Comparison: Placebo vs 300 mg DAC HYP; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Negative Binomial Regression; adjusted for baseline number of T2 lesions; Percent Reduction = 78.73, 95% CI 2-sided [71.33 to 84.22]
Statistical Analysis 2: Comparison: Placebo vs 150 mg DAC HYP; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Negative Binomial Regression; adjusted for baseline number of T2 lesions; Percent Reduction = 70.23, 95% CI 2-sided [59.94 to 77.88]

4. Secondary Outcome: Proportion of Participants Who Relapsed at Week 52
Description: Estimated cumulative proportion of participants relapsed at Week 52, based on the Kaplan-Meier product limit method. Only relapses confirmed by the Independent Neurology Evaluation Committee were included in the analysis.
Time Frame: Week 52
Population: Intent to treat population: all randomized subjects who received at least 1 dose of study medication (excluding 21 subjects from a single site due to a protocol violation in dosing). Participants who did not experience a relapse prior to switching to alternative MS medications or withdrawal from study were censored.
Measure: Number; unit: proportion of participants
Arm/Group | Placebo | 150 mg DAC HYP | 300 mg DAC HYP
Number analyzed (Participants) | 196 | 201 | 203
proportion of participants | 0.36 | 0.19 | 0.20
Statistical Analysis 1: Comparison: Placebo vs 300 mg DAC HYP; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0003, Cox Proportional Hazard — Covariates included were number of relapses in the 1 year prior to study entry (p=0.001), baseline Expanded Disability Status Scale (<=2.5 versus >2.5, p=0.449), and age (<=35 versus >35, p=0.026); Hazard Ratio = 0.49, 95% CI 2-sided [0.33 to 0.72]
Statistical Analysis 2: Comparison: Placebo vs 150 mg DAC HYP; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cox Proportional Hazard — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.30 to 0.67]

5. Secondary Outcome: Mean Change From Baseline in Multiple Sclerosis Impact Scale (MSIS)-29 Physical Impact Score at Week 52
Description: The 29-item Multiple Sclerosis Impact Scale (MSIS-29) is a disease specific patient-reported outcome measure that has been developed and validated to examine the physical and psychological impact of MS from a patient's perspective; it measures 20 physical items and 9 psychological items. Responses use a 5 point Likert scale range from 1 to 5. All questions are to be answered. The total score is the sum of points for all 29 questions, with a minimum score of 29, and a maximum score of 145. A lower total score indicates less physically-related impact while a higher total score indicates greater physically-related impact on a subject's functioning.
Time Frame: Baseline and Week 52
Population: Intent to treat population: all randomized subjects who received at least 1 dose of study medication (excluding 21 subjects from a single site due to a protocol violation in dosing).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 150 mg DAC HYP | 300 mg DAC HYP
Number analyzed (Participants) | 196 | 201 | 203
units on a scale | 3.0 (13.52) | -1.0 (11.80) | 1.4 (13.53)
Statistical Analysis 1: Comparison: Placebo vs 300 mg DAC HYP; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1284, Analysis of Variance — Analysis of variance for difference between treatment groups, controlling for baseline score; Relative Mean Change = -1.93, 95% CI 2-sided [-4.42 to 0.56]
Statistical Analysis 2: Comparison: Placebo vs 150 mg DAC HYP; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0008, Analysis of Variance; Analysis of variance for difference between treatment groups, controlling for baseline score; Relative Mean Change = -4.27, 95% CI 2-sided [-6.76 to -1.78]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the Screening Visit (≤ 21 Days prior to Baseline) through the Follow-Up Visit (Week 72 ± 5 days) or early discontinuation.
Groups:
- Total Active: 150 mg or 300 mg DAC HYP administered as 3 SC injections every 4 weeks for up to 52 weeks
Arm/Group | Placebo | 150 mg DAC HYP | 300 mg DAC HYP | Total Active
Serious Adverse Events (participants affected / at risk) | 53/204 | 32/208 | 36/209 | 68/417
Other Adverse Events (participants affected / at risk) | 128/204 | 109/208 | 111/209 | 220/417
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=204) | 150 mg DAC HYP (N=208) | 300 mg DAC HYP (N=209) | Total Active (N=417)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 1
Diabetes insipidus (Endocrine disorders) | 1 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1
Chronic Hepatitis B (Infections and infestations) | 0 | 1 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1 | 1
Psoas abscess (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 1
Yersinia infection (Infections and infestations) | 0 | 0 | 1 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1 | 1
Multiple sclerosis relapse (Nervous system disorders) | 44 | 19 | 18 | 37
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Temporal lobe epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Ovarian disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=204) | 150 mg DAC HYP (N=208) | 300 mg DAC HYP (N=209) | Total Active (N=417)
Pyrexia (General disorders) | 2 | 7 | 15 | 22
Influenza (Infections and infestations) | 11 | 5 | 12 | 17
Nasopharyngitis (Infections and infestations) | 31 | 30 | 30 | 60
Oral herpes (Infections and infestations) | 10 | 10 | 13 | 23
Pharyngitis (Infections and infestations) | 9 | 13 | 13 | 26
Respiratory tract infection (Infections and infestations) | 11 | 7 | 13 | 20
Upper respiratory tract infection (Infections and infestations) | 14 | 18 | 22 | 40
Alanine aminotransferase increased (Investigations) | 4 | 9 | 12 | 21
Headache (Nervous system disorders) | 21 | 20 | 20 | 40
Multiple sclerosis relapse (Nervous system disorders) | 73 | 45 | 38 | 83
Depression (Psychiatric disorders) | 3 | 10 | 12 | 22
Rash (Skin and subcutaneous tissue disorders) | 6 | 11 | 11 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.